CLINICAL TRIAL: NCT06836063
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Trial to Evaluate Efficacy and Safety of Ropanicant in Patients With Major Depressive Disorder
Brief Title: Study to Evaluate Efficacy and Safety of Ropanicant in MDD Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suven Life Sciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTP2S2911A4B2
Record Dates: First submitted 2025-02-18; First posted 2025-02-20 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: SUVN-911; α4β2; Ropanicant; MDD
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ropanicant Dose Level 1 (Experimental)
  Interventions: Drug: Ropanicant
- Ropanicant Dose Level 2 (Experimental)
  Interventions: Drug: Ropanicant
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ropanicant — Tablet dosage form, twice a day
  Other Names: SUVN-911
  Arms: Ropanicant Dose Level 1; Ropanicant Dose Level 2
Drug: Placebo — Matching placebo tablets, twice a day
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the efficacy of Ropanicant at two different dosage levels compared to placebo in patients with Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
This is a Phase 2b, randomized, double-blind, placebo-controlled, parallel-group, multicenter trial to evaluate the efficacy and safety of Ropanicant versus placebo in patients with MDD. The study will be conducted at multiple centers located in the US.

This study consists of a 4-weeks screening period, 6-weeks treatment period, and a 2-weeks follow-up period. Approximately 195 patients will be randomly assigned to receive Ropanicant Dose Level 1 bid or Dose Level 2 bid, or placebo bid for 6 weeks in a ratio of 1:1:1 (65 patients in each treatment group).

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR) criteria for MDD without psychotic features based on the Mini International Neuropsychiatric Interview (MINI) with a current major depressive episode of at least 4 weeks of duration but no longer than 12 months.
* Patients must have a Clinical Global Impression-Severity (CGI-S) score of ≥4.
* Patients must have a Structured Interview Guide for the Hamilton Depression Rating Scale (SIGH-D) score of ≥20.
* Patients must have a Snaith-Hamilton Pleasure Scale (SHAPS) score of ≥20.
* Patients must have vision and hearing (corrected if needed) sufficient to comply with the testing procedures.

Exclusion Criteria:

* Patients who meet criteria for treatment-resistant depression (TRD) during the current major depressive episode, which is defined as being nonresponders (<50% of symptom improvement) to 2 or more depression treatment periods of adequate dose and duration.
* Patients not in good general health with clinically significant abnormalities as assessed by the investigator and determined by physical examination results, neurological examination results, ECG results, or laboratory assessments.
* Female patients who are pregnant, planning to become pregnant during the study or within 30 days after the last administration of study drug, or breastfeeding.
* Patients with bradycardia (<50 bpm) or tachycardia (>100 bpm) on the ECG results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) total score at Week 6 | Baseline to Week 6
  The MADRS is a clinician-rated scale to assess depressive symptoms which consists from 10 items. The time frame for this scale is the past 7 days. Each item is scored on 7-point scale (0 [absence of symptoms] to 6 [severe]). The total score is the sum of 10 items and can take range from 0 to 60. A higher score represents a higher severity of the level of depression.

SECONDARY OUTCOMES:
Change from Baseline in Clinical Global Impression-Severity (CGI-S) score at Week 6 | Baseline to Week 6
  The CGI-S will be used to rate the severity of each patient's illness related to depressive symptoms on a 7-point scale, which includes the following gradations: 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill.

OTHER OUTCOMES:
Change from Baseline in Snaith-Hamilton Pleasure Scale (SHAPS) score at Week 6 | Baseline to Week 6
  The SHAPS is a subject self- administered scale to measure hedonic capacity which consists of 14 items (total scores range from 14 to 56). Each item has a set of 4 possible responses (Strongly or Definitely Agree, Agree, Disagree and Strongly Disagree). A total score is derived by summing the responses to each item. A higher score represents a higher level of anhedonia.

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Woodland International Research Group LLC, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - Advanced Research Center, Inc., Anaheim, California
  - ProScience Research Group, Culver City, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Synergy San Diego, Lemon Grove, California
  - Excell Research, Inc., Oceanside, California
  - ATP Clinical Research, Orange, California
  - Collaborative Neuroscience Research, Torrance, California
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Premier Clinical Research Institute, Inc, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Panhandle Research and Medical Clinic LLC, Pensacola, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - CenExcel iResearch LLC, Decatur, Georgia
  - CenExcel iResearch LLC, Savannah, Georgia
  - Chicago Research Center Inc., Chicago, Illinois
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - Midwest Research Group, Saint Charles, Missouri
  - Redbird Research, LLC, Las Vegas, Nevada
  - Vector Clinical Trials, Las Vegas, Nevada
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Hassman Research Institue, Marlton, New Jersey
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Neurobehavioral Research Inc., Cedarhurst, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Eximia Research-NC, LLC, Raleigh, North Carolina
  - Sooner Clinical Research, Inc, Oklahoma City, Oklahoma
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - Community Clinical Research, Inc., Austin, Texas
  - North Texas Clinical Trials, LLC, Fort Worth, Texas
  - Memorial Hermann Village, Houston, Texas
  - Core Clinical Research, Everett, Washington